CLINICAL TRIAL: NCT03054363
Title: Phase IB/II Open-label Single Arm Study to Evaluate Safety and Efficacy of Tucatinib in Combination With Palbociclib and Letrozole in Subjects With Hormone Receptor Positive and HER2-positive Metastatic Breast Cancer
Brief Title: Tucatinib, Palbociclib and Letrozole in Metastatic Hormone Receptor Positive and HER2-positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pfizer (Industry); Cascadian Therapeutics Inc. (Industry); Criterium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1661.cc; NCI-2017-01776 (Other: CTRP)
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Tucatinib; Palbociclib; Letrozole; HR-positive; HER2-positive; ER-positive; PR-positive; HER2-targeted therapy; CDK4/6 inhibitor; ONT-380; Ibrance
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1b (Experimental): Tucatinib 300 mg PO BID, palbociclib 125 mg PO daily 21 days on and 7 days off, and letrozole 2.5 mg PO daily on a 28 day cycle length.
  Interventions: Drug: Tucatinib in Combination with Palbociclib and Letrozole
- Phase II (Experimental): Tucatinib 300 mg BID; palbociclib 75 mg PO daily 21 days on, 7 days off; letrozole 2.5 mg PO daily.
  Interventions: Drug: Tucatinib in Combination with Palbociclib and Letrozole

INTERVENTIONS:
Drug: Tucatinib in Combination with Palbociclib and Letrozole — Starting dose of combination therapy :
  Tucatinib 300 mg PO BID Palbociclib 125 mg PO daily 21 day on, 7 days off Letrozole 2.5 mg PO daily
  Other Names: ONT-380; IBRANCE; Femara
  Arms: Phase 1b
Drug: Tucatinib in Combination with Palbociclib and Letrozole — Subjects Tucatinib 300 mg PO BID Palbociclib 75mg PO daily 21 days on followed by 7 days off Letrozole 2.5 mg PO daily.
  Other Names: ONT-380; IBRANCE; Femara
  Arms: Phase II

SUMMARY:
This is a multicenter run-in phase Ib / roll-over phase II study of triple targeted drug combination (HER2-targeted small molecule inhibitor tucatinib, CDK4/6 inhibitor palbociclib and aromatase inhibitor letrozole) as a first or second line of therapy in patients with metastatic hormone receptor positive and HER2-positive breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, single arm, open-label, run-in phase Ib / roll-over phase II study of novel HER2-targeted tyrosine kinase inhibitor tucatinib in combination with CDK4/6 inhibitor palbociclib and aromatase inhibitor letrozole in subjects with HR+/HER2+ locally advanced unresectable or metastatic breast cancer. The study will enroll post-menopausal women and premenopausal women if on treatment with or willing to be treated with standard ovarian suppression. The phase Ib part of the study will determine safety and tolerability of the combination of tucatinib, palbociclib and letrozole to confirm that current RP2D of tucatinib and FDA approved dosing of palbociclib remains the same in the triplet combination. The dose of letrozole will be constant through the study period. Once the safety of the combination is established, we will move to the phase II part of the study in the expansion cohort of subjects at RP2D for the purpose of assessing efficacy while further refining assessment of safety of the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed diagnosis of HR+/HER2+ locally advanced unresectable or metastatic breast cancer. Estrogen or progesterone receptor positivity is defined by IHC according to the most recent ASCO/CAP guidelines. HER2 positivity is defined by standard of care fluorescence in situ hybridization (FISH) and/or 3+ staining by IHC according to the most recent ASCO/CAP guidelines.
2. Measurable and/or evaluable disease per RECIST 1.1 criteria and/or RANO-BM criteria

   . Bone only disease is allowed.
3. CNS inclusion criteria:

   * Subjects without CNS metastases are eligible. Note: brain imaging is not required for asymptomatic subjects without known brain metastatic disease prior to enrollment into the study
   * Subjects with untreated asymptomatic CNS metastases not needing immediate local therapy in the opinion of investigator are eligible. For subjects with untreated asymptomatic CNS lesions > 2.0 cm by contrast-enhanced MRI, discussion with and approval from the Lead PI is required prior to enrollment
   * Subjects with stable brain metastases previously treated with radiation therapy or surgery are allowed to enroll, provided that they are off corticosteroids or on stable/tapering dose of corticosteroids and stability of CNS metastatic disease for at least 4 weeks has been demonstrated, with the last MRI taken within 2 weeks prior to cycle 1 day 1 of the study.

   Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions
4. Age ≥ 18 years
5. ECOG performance status 0-1
6. Life expectancy of more than 6 months, in the opinion of the investigator
7. Study subjects should be post-menopausal women; premenopausal women are eligible if on ovarian suppression, or agreeable to mandatory ovarian suppression. Women of childbearing potential, defined as premenopausal women who are not permanently sterile (i.e., due to hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or bilateral tubal occlusion) are required to have negative pregnancy tests prior to initiation of treatment.
8. Prior treatments:

   * Subjects should have received at least two approved HER2-targeted agents (trastuzumab, pertuzumab, or TDM-1) in the course of their disease
   * Subjects should have had at least 1 line of prior HER2-targeted therapy in the metastatic setting, with the exception of asymptomatic subjects with oligometastatic or bone / soft tissue only disease who, on investigator opinion, are appropriate for a single agent antiendocrine therapy per NCCN guidelines
   * Subjects who have had up to 2 lines of prior endocrine therapy in the metastatic setting are allowed. Prior adjuvant and/or neoadjuvant endocrine regimens are allowed and not counted towards this limit
9. Adequate organ and marrow function as defined below:

   * Absolute neutrophil count ≥ 1,500/mm3
   * Platelets ≥ 75,000/mm3
   * Hemoglobin ≥ 9.0 mg/dL without red blood cell transfusion ≤ 7 days prior to Cycle 1Day 1 of therapy
   * Total serum bilirubin ≤ 1.5 X upper limit of normal (ULN) except for subjects with known Gilbert's disease, who may enroll if the conjugated bilirubin is ≤ 1.5 ULN
   * AST (SGOT)/ALT (SGPT) ≤2.5 X ULN;
   * Serum creatinine ≤ 1.5 mg/dL
   * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 X ULN unless on medication known to alter INR and aPTT
   * Left ventricular ejection fraction (LVEF) ≥ 50% (as assessed by ECHO or MUGA) documented within 4 weeks prior to first dose of study treatment
   * Serum or urine pregnancy test (for women of childbearing potential) negative ≤ 7 days of starting treatment
10. Ability to understand and the willingness to sign a written informed consent and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
11. Subject or legally authorized representative of a subject must provide signed informed consent per a consent document that has been approved by an institutional review board or independent ethics committee (IRB/IEC) prior to initiation of any study-related tests or procedures that are not part of standard-of-care for the subject's disease.

Exclusion criteria:

1. Subjects with previously treated progressing brain metastases are excluded from the study
2. Subjects with known brain metastases and contraindications to undergo contrast MRI imaging of the brain are excluded from the study
3. Pregnancy or breast feeding
4. Current active treatment with an investigational agent
5. Known history of hypersensitivity to aromatase-inhibitor drugs
6. Any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the exception of peripheral neuropathy, which must have resolved to ≤ Grade 2, and alopecia
7. Previous treatment with lapatinib, neratinib, afatinib, or other investigational EGFR-family receptor tyrosine kinase inhibitor or HER2 tyrosine kinase inhibitor
8. Previous treatment with palbociclib, abemaciclib, ribociclib or other investigational CDK4/6 inhibitors
9. Any systemic anti-cancer therapy (including hormonal therapy), radiation, or experimental agent ≤ 2 weeks of first dose of study treatment
10. Active bacterial, fungal or viral infections requiring treatment with IV antibiotic, IV antifungal, or IV anti-viral drugs
11. Known hepatitis B (HBV), hepatitis C (HCV) or human immunodeficiency virus (HIV) infections. Note: pretesting is not required.
12. Inability to swallow pills or any significant gastrointestinal disease which would preclude the adequate oral absorption of medications
13. Use of prohibited medications within 3 elimination half-lives prior to first dose of the study treatment
14. Known myocardial infarction, severe/unstable angina, percutaneous transluminal coronary angioplasty/stenting (PTCA), or coronary artery bypass graft (CABG) within 6 month of the first dose of the study treatment
15. Clinically significant cardio-vascular disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension (defined as persistent systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications), or any history of symptomatic congestive heart failure (CHF)
16. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the subject inappropriate for entry into the study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Shagisultanova, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Arizona, Tucson, Arizona
  - University of Colorado Denver, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Stony Brook University, Stony Brook, New York
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shagisultanova E, Crump LS, Borakove M, Hall JK, Rasti AR, Harrison BA, Kabos P, Lyons TR, Borges VF. Triple Targeting of Breast Tumors Driven by Hormonal Receptors and HER2. Mol Cancer Ther. 2022 Jan;21(1):48-57. doi: 10.1158/1535-7163.MCT-21-0098. Epub 2021 Nov 2. PMID 34728571
- [Derived] Shagisultanova E, Gradishar W, Brown-Glaberman U, Chalasani P, Brenner AJ, Stopeck A, Parris H, Gao D, McSpadden T, Mayordomo J, Diamond JR, Kabos P, Borges VF. Safety and Efficacy of Tucatinib, Letrozole, and Palbociclib in Patients with Previously Treated HR+/HER2+ Breast Cancer. Clin Cancer Res. 2023 Dec 15;29(24):5021-5030. doi: 10.1158/1078-0432.CCR-23-0117. PMID 37363965

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b: Tucatinib in Combination with Palbociclib and Letrozole (Safety Cohort): Starting dose of combination therapy :
  Tucatinib 300 mg PO BID Palbociclib 125 mg PO daily 21 day on, 7 days off Letrozole 2.5 mg PO daily
- Phase II: The study completed the final phase Ib safety analysis on January 31, 2019. Tucatinib 300 mg BID; palbociclib 75 mg PO daily 21 days on, 7 days off; letrozole 2.5 mg PO daily..
Period: Overall Study
Arm/Group | Phase 1b | Phase II
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase Ib: Tucatinib 300 mg PO BID Ppalbociclib 125 mg PO daily 21 days on and 7 days off Letrozole 2.5 mg PO daily on a 28 day cycle length.
- Phase II: Tucatinib 300 mg PO BID Palbociclib 75mg PO daily 21 days on followed by 7 days off Letrozole 2.5 mg PO daily.
- Total: Total of all reporting groups
Arm/Group | Phase Ib | Phase II | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.55) | 53.12 (15.49) | 51.91 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 18 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib Primary Outcome: Proportion of Patients Who Experienced DLTs Attributable to Palbociclib, Tucatinib, or Both
Description: To measure safety and tolerability of tucatinib used in combination with palbociclib and letrozole, we will assess the proportion of subjects experiencing dose-limiting toxicities (DLTs) potentially attributable to tucatinib, palbociclib, or both drugs, and compare them to predefined safety thresholds. DLT was defined as any grade ≥ 3 nonhematologic adverse event, grade 3 neutropenia with fever, grade 3 thrombocytopenia with bleeding, or any hematologic toxicity grade ≥ 4 using NCI CTCAE version 4.03. Safety was considered clinically meaningfully altered if ≥60% of subjects experienced DLTs secondary palbociclib, ≥20% of subjects had toxicity secondary to tucatinib, or ≥50% of subjects had DLTs attributable to both drugs. If the proportion of patients with DLTs cross safety boundaries, doses of tucatinib, palbociclib or both medications would be decreased. Letrozole dose was kept constant for all study subjects.
Time Frame: 15 months (From date of first consent until final safety analysis of Phase Ib)
Population: Among the 20 phase Ib patients, 1 (5%) had a dose reduction of tucatinib, and 9 (45%) had a dose reduction of palbociclib for DLTs. Two patients (10%) discontinued palbociclib because of DLTs (neutropenia) and continued tucatinib and letrozole. One patient (5%) discontinued letrozole for toxicity, and continued tucatinib and palbociclib. The pre-defined safety boundaries were not crossed.
Measure: Number; unit: percentage of participants
Groups:
- Baseline Starting Dose Patients for Phase Ib (Tucatinib 300mg, Palbociclib 125mg, Letrozole 2.5mg): Enroll 10 subjects at the baseline starting doses (DL1) of tucatinib 300 mg PO BID, palbociclib 125 mg PO daily 21 days on and 7 days off, and letrozole 2.5 mg PO daily on a 28 day cycle length. After 10 subjects are accrued to the study and complete at least 1 cycle of treatment, an interim analysis of the safety phase Ib cohort will be done.
  Plan - 10 subjects enrolled, completed at least one cycle of treatment (28 days) and evaluable for safety analysis: If there are 7 or fewer subjects experience DLTs due to palbociclib, 3 or fewer subjects experience DLTs due to tucatinib, and 7 or fewer subjects experience DLTs potentially attributable to both drugs, then the interim safety of the Phase Ib cohort will be considered acceptable and accrual will continue to enroll to 20 subjects without change of the starting doses.
  Tucatinib in Combination with Palbociclib and Letrozole (Safety Cohort): Starting dose of combination therapy :
  Tucatinib 300 mg PO BID Palbociclib 125 mg PO daily 21 day on, 7 days off Letrozole 2.5 mg PO daily
- Dose-reduced Patients for Phase II (Tucatinib 300mg, Palbociclib 75mg, Letrozole 2.5mg): Patients who participated in the phase Ib part of the study and continued into the phase II part and had their palbociclib dose reduced.
- Overall Patient Cohort: All patients from both parts of the study.
Arm/Group | Baseline Starting Dose Patients for Phase Ib (Tucatinib 300mg, Palbociclib 125mg, Letrozole 2.5mg) | Dose-reduced Patients for Phase II (Tucatinib 300mg, Palbociclib 75mg, Letrozole 2.5mg) | Overall Patient Cohort
Number analyzed (Participants) | 20 | 13 | 20
percentage of participants | 100 | 65 | 100

2. Primary Outcome: Phase II Primary Outcome: Median Progression-free Survival (mPFS)
Description: To measure efficacy of tucatinib used in combination with palbociclib and letrozole, the median PFS (primary objective of Phase II) will be assessed. mPFS is defined as the time from allocation to the first documented disease progression according to RECIST 1.1, or death due to any cause, whichever occurs first. For subjects with brain metastatic disease enrolled in the study, assessment of bi-compartmental mPFS in the non-CNS and CNS compartments, defined as the time from allocation to the first documented disease progression according to RECIST 1.1 and/or RANO-BM criteria, or death due to any cause, whichever occurs first.
  For patient with CNS metastases who had an event of isolated CNS progression, underwent local therapy, and remained on study per protocol, mPFS was calculated as the time from the start of treatment until the first CNS progression.
Time Frame: 4 years (data cutoff of PFS calculation was when PFS became mature according to study statistician)
Population: There were 40 evaluable patients for this efficacy outcome. Two patients were non-evaluable because they received less than 2 cycles of treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Overall Patient Cohort: All response-evaluable patients from the Phase Ib or Phase II part of the study. Evaluable patients received at least 2 cycles of treatment and one radiographic tumor assessment.
- CNS Cohort: Response-evaluable patients with CNS metastases.
- Non-CNS Cohort: Response-evaluable without CNS metastases.
Arm/Group | Overall Patient Cohort | CNS Cohort | Non-CNS Cohort
Number analyzed (Participants) | 40 | 15 | 25
months | 8.4 [6.6 to 10.8] | 8.2 [5.4 to 20.1] | 10.0 [7.2 to 14.9]

3. Secondary Outcome: Phase Ib Secondary Outcome: Tucatinib and Palbociclib AUC[0-6] Post Tucatinib and Palbociclib Dose
Description: Pharmacokinetic (PK) assessments of blood levels of tucatinib and palbociclib will be performed on Cycle 1 Day 15 and Cycle 2 Day 1 of therapy in 20 participants enrolled in the phase Ib part of the study. Plasma samples will be collected to measure levels of tucatinib and its hydroxyl metabolite ONT-993, as well as levels of palbociclib and, if needed, its metabolites at steady state on Cycle 1 Day 15. The area under the curve (AUC) of the concentration vs. time plot is computed from 0 to 6 hours after the tucatinib and palbociclib dose.
Time Frame: 0, 0.5, 1, 2, 3, 4, and 6 hours post-dose
Population: All 20 patients enrolled in Phase Ib were included in PK analysis.
Measure: Mean (Full Range); unit: h*ng/mL
Groups:
- Baseline Starting Dose Patients (1-20): Tucatinib in Combination With Palbociclib and Letrozole: Enroll 10 subjects at the baseline starting doses (DL1) of tucatinib 300 mg PO BID, palbociclib 125 mg PO daily 21 days on and 7 days off, and letrozole 2.5 mg PO daily on a 28 day cycle length. After 10 subjects are accrued to the study and complete at least 1 cycle of treatment, an interim analysis of the safety phase Ib cohort will be done.
  Plan - 10 subjects enrolled, completed at least one cycle of treatment (28 days) and evaluable for safety analysis: If there are 7 or fewer subjects experience DLTs due to palbociclib, 3 or fewer subjects experience DLTs due to tucatinib, and 7 or fewer subjects experience DLTs potentially attributable to both drugs, then the interim safety of the Phase Ib cohort will be considered acceptable and accrual will continue to enroll to 20 subjects without change of the starting doses.
  Tucatinib in Combination with Palbociclib and Letrozole (Safety Cohort): Starting dose of combination therapy :
  Tucatinib 300 mg PO BID Palbociclib 125 mg PO daily 21 day on, 7 days off Letrozole 2.5 mg PO daily
Arm/Group | Baseline Starting Dose Patients (1-20): Tucatinib in Combination With Palbociclib and Letrozole
Number analyzed (Participants) | 20
h*ng/mL
  Palbociclib | 647 [183.6 to 1983]
  Tucatinib | 2433 [1289 to 4022]
  ONT-993 (Tucatinib metabolite) | 340 [156.5 to 943.1]

4. Secondary Outcome: Phase II Secondary Outcome: Palbociclib AUC[10-19] Post Tucatinib and Palbociclib Dose
Description: Additional pharmacokinetic (PK) assessment will be done in 5 to 10 patients enrolled in phase II part of the study to evaluate the levels of tucatinib and palbociclib. These PKs will be done on Cycle 1 Day 9 and Cycle 2 Day 9. Prior to the first set of PKs, on Cycle 1 Days 1-8, patient will take palbociclib and letrozole; tucatinib will be on hold. Tucatinib will be started per usual study schedule after the first set of PKs is obtained on Day 9. Prior to the second set of PKs, on Cycle 2 Days 1-8, patient will take palbociclib, letrozole and tucatinib (all study drugs) per usual study schedule. On the day prior to PK evaluation (Day 8 of Cycle 1 and Day 8 of Cycle 2), patient should consume high calorie / high fat meal and take study drugs. On the next day, plasma samples will be collected to measure PKs at 10, 13, 16 and 19 hrs +/- 10 minutes post dose.
Time Frame: 10, 13, 16, and 19 hours post-dose
Population: 9 patients were studied for Phase II PKs.
Measure: Mean (Full Range); unit: h*ng/mL
Groups:
- Overall Patient Cohort: All 9 patients who were evaluated for PK analysis.
Arm/Group | Overall Patient Cohort
Number analyzed (Participants) | 9
h*ng/mL | 656 [506 to 1108]

5. Secondary Outcome: Phase II Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was assessed in patients with measurable lesions and defined as the proportion of patients with complete response, partial response, or stable disease for 6 months or more. It is one of the parameters used to assess tumor response in this study and was evaluated using RECIST 1.1 (and/or RANO-BM for patients with CNS disease).
Time Frame: 4 years
Population: 27 patients of the 40 who were evaluable for safety were analyzable for this tumor response outcome because they had measurable lesions.
Measure: Number; unit: percentage of participants
Groups:
- Patients With Measurable Lesions (n=27): All patients with measurable lesions from either part of the study.
Arm/Group | Patients With Measurable Lesions (n=27)
Number analyzed (Participants) | 27
percentage of participants | 70.4

6. Secondary Outcome: Phase II Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) is defined as the proportion of subjects who had complete or partial response by RECIST 1.1 (and/or RANO-BM for patients with CNS disease).
Time Frame: 4 years
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Measurable Lesions (n=27)
Number analyzed (Participants) | 27
percentage of participants | 44.5

7. Secondary Outcome: Phase II Secondary Outcome: Median Duration of Response (mDOR)
Description: Median duration of response (mDOR) is defined as the time from enrollment in the clinical trial until objective tumor progression or death, whichever occurs first.
Time Frame: 4 years
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Patients With Measurable Lesions (n=27)
Number analyzed (Participants) | 27
months | 13.9 [5.51 to 31.8]

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Groups:
- Phase Ib: Tucatinib 300 mg PO BID, palbociclib 125 mg PO daily 21 days on and 7 days off, and letrozole 2.5 mg PO daily on a 28 day cycle length.
Arm/Group | Phase Ib | Phase II
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 9/20 | 7/22
Other Adverse Events (participants affected / at risk) | 20/20 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib (N=20) | Phase II (N=22)
Sepsis (Infections and infestations) | 1 (1) | 1 (3)
Pleural Effusions, Bilateral (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hydronephrosis with Hydrourters, Bilateral (Renal and urinary disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Upper respiratory infection, possible (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Malnutrition, Severe (General disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
AST Increase (Investigations) | 1 (1) | 0 (0)
ALT Increase (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Thromboembolic Event, Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib (N=20) | Phase II (N=22)
Abdominal Pain (Gastrointestinal disorders) | 5 (10) | 4 (4)
Acne (acneform rash) (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 (4) | 0 (0)
Adenopathy (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (6) | 3 (5)
Alkaline Phosphatase increased (Infections and infestations) | 2 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 7 (16) | 3 (16)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 5 (7)
Arthralgias (Musculoskeletal and connective tissue disorders) | 3 (6) | 4 (7)
Aspartate Aminotransferase Increased (Investigations) | 3 (8) | 3 (4)
Pneumonia, Atypical (Infections and infestations) | 1 (1) | 1 (1)
Pain (General disorders) | 12 (32) | 10 (18)
Tremors, Bilateral hands (Nervous system disorders) | 1 (1) | 1 (1)
Bilirubin, Increased (Investigations) | 2 (3) | 2 (3)
Bloating (Gastrointestinal disorders) | 2 (3) | 0 (0)
Chills (General disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (1)
Neutrophil Count, Decreased (Investigations) | 17 (76) | 16 (79)
Platelet Count Decreased (Investigations) | 6 (23) | 1 (6)
White Blood Cell Count Decreased (Investigations) | 11 (43) | 5 (27)
Diarrhea (Gastrointestinal disorders) | 11 (35) | 16 (30)
Dizziness (Nervous system disorders) | 5 (5) | 5 (8)
Dry Eyes (Eye disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Edema (General disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Numbness (General disorders) | 2 (3) | 0 (0)
Fall (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 13 (20) | 14 (21)
fever (General disorders) | 4 (8) | 3 (3)
Flu like symptoms (General disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 7 (10) | 6 (7)
Hoarseness (General disorders) | 2 (2) | 1 (1)
Hot Flashes (General disorders) | 2 (2) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (9) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (8) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (10) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (7) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Infection (Infections and infestations) | 12 (19) | 6 (7)
Increased INR (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 3 (20) | 3 (12)
maculopapular rash (Skin and subcutaneous tissue disorders) | 2 (8) | 3 (3)
Memory Impairment (Nervous system disorders) | 1 (1) | 1 (1)
Mucositis (Infections and infestations) | 9 (17) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (25) | 12 (18)
Neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Parethesias (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin Laceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6) | 1 (2)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (20) | 6 (11)
Weight Loss (General disorders) | 5 (6) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Dyspepsia/Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Creatinine, Elevated (Investigations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03054363/Prot_SAP_ICF_000.pdf